CLINICAL TRIAL: NCT02355899
Title: Evaluation of the Suitability of PD P 506 A in the Photodynamic Therapy of Distal Subungual Onychomycosis (DSO) of the Great Toenail.
Brief Title: Evaluation of the Suitability of PD P 506 A in the PDT of Distal Subungual Onychomycosis (DSO) of the Great Toenail.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: photonamic GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OM 01
Record Dates: First submitted 2015-01-22; First posted 2015-02-04 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD P 506 A-PDT (Experimental): One PD P 506 A-patch will be administered to each great toenail for 4 hours. After removal of the study medication the study nail(s) s will be illuminated with red light of defined wavelength (PDT).
  Interventions: Drug: PD P 506 A

INTERVENTIONS:
Drug: PD P 506 A — PD P 506 A is a dermal patch of 4 cm² in size loaded with 2 mg 5-ALA (as 5-ALA HCl) per cm².
  Other Names: Alacare®

SUMMARY:
This study evaluates the potential usefulness of photodynamic therapy with PD P 506 A in patients with distal subungual onychomycosis of the great toenail. Patients will receive four PDT treatments with PD P 506 A in weekly intervals.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 - 75 years of age
* Females up to an age of 75 years provided that they are postmenopausal, i.e. with spontaneous amenorrhea for at least 12 months or not of childbearing potential because of tubal ligation or hysterectomy
* DSO of at least one of the great toe(s) affecting 20% to 60% of the target nail without spikes, confirmed before Visit 1 by at least one of the three methods: the methods of KOH test, periodic acid-Schiff (PAS) stain and mycology culture
* The toenail infection can be due to a dermatophyte, yeast or mixed infections (dermatophyte and non-dermatophyte)
* Toenails have to be cut regularly (indicator for existing growth)
* Signed written informed consent

Exclusion Criteria:

* Patients with the target toenail involving the matrix (lunula) or having less than 2 mm clear (unaffected) nail plate length beyond the proximal fold
* Presence of dermatophytoma (defined as demarcated and localised thick masses (≥ 3 mm) of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the target nail
* Other conditions than DSO known to cause abnormal nail appearance
* Topical antifungal treatment of the nails within 1 month before PDT
* Systemic use of antifungal treatment within 3 months before PDT
* Patients who are unwilling to provide nail clippings
* Patients who have been previously reported to be allergic against 5-aminolevulinic acid or other ingredients of PD P 506 A
* Diagnosis of porphyria
* Diagnosis of polyneuropathy
* Dementia or psychic condition that might interfere with the ability to understand the study and thus give written informed consent
* Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Percentage of nails with Clinically Complete Cure | 12 months after last study treatment
  The Complete Clinical Clearance of each treated nail will be determined 3, 6 and 12 months after last study treatment. Based on a visual inspection, the nail(s) will either be defined as "completely cleared" or "partially" or "not cleared".
  To be defined as "completely cleared", a nail must show 100% absence of the 4 following clinical signs of onychomycosis (according to Scher et al., J Am Acad Dermatol. 2007 Jun;56(6):939-44):
  * Residual changes of the nail plate compatible with dermatophyte infection
  * White/yellow or orange brown/patches or streaks in or beneath the nail
  * Lateral onycholysis with debris in an otherwise clear nail plate
  * Hyperkeratoses on the lateral nail plate/nailfold edge. If the nail shows an improvement but still one of the above signs, it will be rated as "partially cleared".
  If the nail shows no improvement in comparison to the Screening Visit, it will be rated as "not cleared".

SECONDARY OUTCOMES:
Percentage of nails with negative laboratory test results for onychomycosis (KOH test, periodic acid-Schiff (PAS) stain and mycology culture). | 12 months after last study treatment
Percentage of nails with Clinically Complete Cure | 3 and 6 months after last study treatment
  The Complete Clinical Clearance of each treated nail will be determined 3, 6 and 12 months after last study treatment. Based on a visual inspection, the nail(s) will either be defined as "completely cleared" or "partially" or "not cleared".
  To be defined as "completely cleared", a nail must show 100% absence of the 4 following clinical signs of onychomycosis (according to Scher et al., J Am Acad Dermatol. 2007 Jun;56(6):939-44):
  * Residual changes of the nail plate compatible with dermatophyte infection
  * White/yellow or orange brown/patches or streaks in or beneath the nail
  * Lateral onycholysis with debris in an otherwise clear nail plate
  * Hyperkeratoses on the lateral nail plate/nailfold edge. If the nail shows an improvement but still one of the above signs, it will be rated as "partially cleared".
  If the nail shows no improvement in comparison to the Screening Visit, it will be rated as "not cleared".
Frequency of adverse events | During the treatment phase on day 0, 7, 14 and 21, and 3, 6 and 12 months after last study treatment
Severity (grade1-5) of adverse events | During the treatment phase on day 0, 7, 14 and 21, and 3, 6 and 12 months after last study treatment
  The severity of AEs is defined as:
  * Grade 1 = mild
  * Grade 2 = moderate
  * Grade 3 = severe
  * Grade 4 = life-threatening
  * Grade 5 = fatal
Frequency of local reactions. | During the treatment phase on day 0, 7, 14 and 21, and 3, 6 and 12 months after last study treatment
  Photodynamic therapy is intended to produce a phototoxic reaction, which is part of the desired effect. After PDT, treated toes may show local reactions such as redness and swelling.
Severity (grade1-3) of local reactions. | During the treatment phase on day 0, 7, 14 and 21, and 3, 6 and 12 months after last study treatment
  The severity of local reactions is defined as:
  * Grade 1 = mild
  * Grade 2 = moderate
  * Grade 3 = severe
One photo of each treated toenail at the beginning of each visit | At screening visit (up to 4 weeks before first treatment), during the treatment phase on day 0, 7, 14 and 21, and 3, 6 and 12 months after last study treatment.
  Documentation of the course of the study for each treated toenail.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf-Markus Szeimies, Prof. Dr., Principal Investigator — KLINIKUM VEST GMBH Knappschaftskrankenhaus Recklinghausen
Locations (2):
- Germany (2):
  - Klinik für Dermatologie, Klinikum Lippe, Detmold
  - Klinik für Dermatologie und Allergologie KLINIKUM VEST GMBH Knappschaftskrankenhaus Recklinghausen, Recklinghausen

IPD SHARING:
Plan to Share IPD: No